CLINICAL TRIAL: NCT05461053
Title: A Randomized Controlled Trial for Conservative Management of Cutaneous Abscess Using Topical Anesthetic in Children as Compared to Standard Management
Brief Title: Conservative Management of Cutaneous Abscess
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21120103
Record Dates: First submitted 2022-07-06; First posted 2022-07-15 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cutaneous Abscess
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Warm Compress application (No Intervention): The control group will receive instructions on applying warm compresses, the current standard of care. The patient or parent/guardian will be directed to apply a warm compress to the abscess or soak the area in warm water for 15 minutes. The application/soak will be done 4 times during the day.
- LMX4-A topical anesthetic application (Experimental): The intervention group will be prescribed a course of LMX4 with application of a non-permeable dressing (Tegaderm, 3M, St Paul, MN) until time of spontaneous drainage, treatment failure, or resolve of pain. LMX4 is a topical anesthetic consisting of 4% lidocaine which is Food and Drug Administration (FDA) approved for topical use in children.
  Interventions: Drug: LMX 4 Topical Cream

INTERVENTIONS:
Drug: LMX 4 Topical Cream — The intervention group will be prescribed a course of LMX4 with application of a non-permeable dressing (Tegaderm, 3M, St Paul, MN) until time of spontaneous drainage, treatment failure, or resolve of pain. LMX4 is a topical anesthetic consisting of 4% lidocaine which is Food and Drug Administration (FDA) approved for topical use in children.
  Other Names: lidocaine
  Arms: LMX4-A topical anesthetic application

SUMMARY:
This is a single center non-blinded randomized trial of topical anesthetic cream to usual care (warm compresses and time) for superficial, non-perianal abscesses in children under 18 years of age. The primary outcome is time to spontaneous drainage. The secondary outcomes are return to emergency room/hospital/care provider and need for incision and drainage. Information on patient experience using standardized patient reported outcome measures for health-related quality of life will also be gathered. The findings of this study will provide more robust evidence of the benefit of this treatment including a potential reduction in cost and allow for more widespread dissemination.

DETAILED DESCRIPTION:
Cutaneous abscesses are a common problem in the pediatric population, leading to a substantial number of emergency room and primary care visits each year. Historically, treatment consisted of antibiotics and surgical drainage, but as our understanding of these disease processes has progressed, treatment has moved away from invasive drainage procedures except when necessary. Now, most patients are treated with warm compresses or warm baths to the area until spontaneous resolution occurs. Recent data has demonstrated that the application of topical anesthetic cream to a cutaneous abscess underneath a non-permeable dressing can lead to improved rates of spontaneous drainage. Although this method is being used with success at our institution, its true benefit is unknown, preventing widespread dissemination of the practice. We are therefore proposing a prospective trial to evaluate the benefit of this treatment on pediatric patients. This is a single center non-blinded randomized trial of topical anesthetic cream to usual care (warm compresses and time) for superficial, non-perianal abscesses in children under 18 years of age. The primary outcome is time to spontaneous drainage. The secondary outcomes are return to emergency room/hospital/care provider and need for incision and drainage. Information on patient experience using standardized patient reported outcome measures for health-related quality of life will also be gathered. The findings of this study will provide more robust evidence of the benefit of this treatment including a potential reduction in cost and allow for more widespread dissemination.

ELIGIBILITY:
Inclusion Criteria:

* <18 years of age
* Single, localized soft tissue abscess <3 cm in size by clinical or imaging criteria

Exclusion Criteria:

* Signs of systemic illness/infection including but not limited to temperature > 100.4, lethargy, or poor oral intake;
* A decision by an attending physician that incision and drainage is necessary;
* Inpatient admission; immunocompromised patients; soft tissue abscesses involving the perineum (labia, scrotum, penis, perianal), hands/feet, or face;
* Previous antibiotic use in the past seven days or previous attempt by a clinician/provider at drainage;
* Current drainage from abscess.
* Lidocaine allergy

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Time to Spontaneous Discharge | Enrollment + 7-14 Days
  Patient/Caregiver will be called to learn date of spontaneous discharge

SECONDARY OUTCOMES:
Rate of Failure | Enrollment + 30 Days
  Study team will review medical records for hospital admission, need for incision and drainage, or additional medication treatment

OTHER OUTCOMES:
Pain Interference PROMIS Pediatric Item Bank v2.0 - Pain Interference - Short Form 8a | Enrollment + 7-14 Days
  PROMIS Pediatric Item Bank v2.0 - Pain Interference - Short Form 8a, range 8-40, lower score better
Pain Interference PROMIS Pediatric Item Bank v2.0 - Pain Interference | Enrollment + 7-14 Days
  PROMIS Pediatric Item Bank v2.0 - Pain Interference, range 20-100, lower score better
Pain Interference PROMIS Parent Proxy Item Bank v2.0 - Pain Interference - Short Form 8a | Enrollment + 7-14 Days
  PROMIS Parent Proxy Item Bank v2.0 - Pain Interference - Short Form 8a, range 8-40, lower score better
Pain Interference PROMIS Parent Proxy Item Bank v2.0 - Pain Interference | Enrollment + 7-14 Days
  PROMIS Parent Proxy Item Bank v2.0 - Pain Interference, range 13-65, lower score better
Global Health PROMIS Pediatric Scale v1.0 - Global Health 7+2 | Enrollment + 7-14 Days
  PROMIS Pediatric Scale v1.0 - Global Health 7+2, range 9-45, lower score better
Global Health PROMIS Parent Proxy Scale v1.0 - Global Health 7+2 | Enrollment + 7-14 Days
  PROMIS Parent Proxy Scale v1.0 - Global Health 7+2, range 9-45, lower score better

CONTACTS AND LOCATIONS:
Overall Officials: Brian Gulack, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States